CLINICAL TRIAL: NCT04787419
Title: The Role of Probiotics in Chronic Cholestasis to Prevent Gastrointestinal Diseases in Pediatric Patients in Cipto Mangunkusumo Hospital
Brief Title: Probiotics in Pediatric Chronic Cholestasis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Fatima Safira Alatas, SpA(K), PhD, Pediatric gastrohepatoenterologist consultant, clinical professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-07-0733
Record Dates: First submitted 2021-02-09; First posted 2021-03-08 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Cholestatic Liver Disease
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both placebo and probiotics have the exact same packaging. batch production numbers are printed, ended with either "0" or "1". code will be revealed by third party (production and packaging team) upon study completion (following data analysis)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotics (Experimental): 2 sachets per day for 4 weeks.
  1 sachet of probiotics (1gram) contains: Viable Counts 1 x 107 CFU/g living bacteria in dual pH dependent release coated (Lactobacillus acidophilus, Bifidobacterium longum, Streptococcus thermophilus), Vitamin C 10 mg, Vitamin B1 0.5 mg, Vitamin B2 0.5 mg, Vitamin B6 0.5 mg, Niacin 2 mg.
  Interventions: Combination Product: probiotics
- placebo (Placebo Comparator): 2 sachets per day for 4 weeks.
  1 sachet of placebo (1gram) contains: saccharum lactis
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — saccharum lactis
  Arms: placebo
Combination Product: probiotics — Lactobacillus acidophilus, Bifidobacterium longum, Strepococcus thermophilus
  Arms: probiotics

SUMMARY:
double blinded RCT (probiotics vs placebo) given to pediatric patients with chronic cholestasis for 4 weeks duration. baseline characteristics (antropometry, gastrointestinal symptoms, laboratory examinations) would be compared pre vs post treatment

DETAILED DESCRIPTION:
In mice model of cirrhosis and ascites, there is an increased intestinal permeability (leaky gut syndrome), subsequently leads to bacterial translocation. Bacterial translocation ultimately leads to bacterial overgrowth and increases associated morbidity, for instance, protracted diarrhea.

This RCT aims to administer probiotics product (lacto-B) in pediatric patients with chronic cholestasis (cholestasis > 4 weeks, evidenced from laboratory examination results).

method: double-blinded RCT

regimen: (identical, plain silver packaging, with code 0/1 --> revealed by 3rd party upon study completion)

intervention group: lacto-B 2 sachet per day for 4 weeks (28 days) each sachet of lacto-B contains: Viable Counts 1 x 107 CFU/g living bacteria in dual pH dependent release coated (Lactobacillus acidophilus, Bifidobacterium longum, Streptococcus thermophilus), Vitamin C 10 mg, Vitamin B1 0.5 mg, Vitamin B2 0.5 mg, Vitamin B6 0.5 mg, Niacin 2 mg.

control group: placebo sachet (saccharum lactis 1gr)

outcomes will be measured following completion of 4 weeks-course of probiotics/placebo

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with chronic cholestasis (>4 weeks evidence of cholestasis from laboratory evidence)
* patient/guardian give consent to participate

Exclusion Criteria:

* immunocompromised
* consumed antibiotic within 2 weeks prior to recruitment time
* patient already consuming probiotic-added formula (any probiotic supplementation or formula milk with added probiotic)

Ages: 29 Days to 215 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
macroscopic fecal analysis | 28th day of product consumption
  consistency of stool according to Bristol stool chart
microscopic fecal erythrocyte count | 28th day of product consumption
  fecal erythrocyte count per high power field
microscopic fecal leukocyte count | 28th day of product consumption
  fecal leukocyte count per high power field
fecal calprotectin | 28th day of product consumption
  fecal calprotectin measured using ELISA technique, reported in micrograms/gram
gut microbiota diversity | 28th day of product consumption
  PCR of gut microbiota diversity
presence of intestinal bacteria overgrowth | 28th day of product consumption
  measured using hydrogen breath test

SECONDARY OUTCOMES:
albumin | 28th day of product consumption
  serum albumin level measured in umol/L
ALT | 28th day of product consumption
  serum ALT measured in u/L
AST | 28th day of product consumption
  serum AST measured in u/L
ALP | 28th day of product consumption
  serum ALP measured in u/L
GGT | 28th day of product consumption
  serum GGT measured in u/L
bilirubin level | 28th day of product consumption
  serum total, direct and indirect bilirubin levels measured in u/L
incidence of diarrhea | day 1- day 28 of product consumption
  any episode of diarrhea within intervention period (>3x/day, loose bowel, or exceeds usual frequency for infants)
antibiotic use | day1 - day 28 of product consumption
  any antibiotic consumption as indicated by presence of infection (any organ system)

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Safira Alatas, MD, PhD, Principal Investigator — Department of Child Health Cipto Mangunkusumo Hospital, Faculty of Medicine Universitas Indonesia
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided